CLINICAL TRIAL: NCT07060898
Title: Radicle Clarity™ 25_RAM: A Randomized, Double-Blind, Placebo-Controlled Direct-to-Consumer Study Assessing the Impact of Health and Wellness Products on Cognitive Function and Related Health Outcomes
Brief Title: Impact of a Novel Brain Longevity Supplement Containing the Postbiotic Urolithin A (Mitopure) on Cognitive Function and Related Health Outcomes
Acronym: CLARITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amazentis SA (Industry)
Collaborators: Radicle Science (sponsor) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: RADX-SP-2506_RAM
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Aging; Cognitive Decline; Brain Fog; Cognitive Function
Keywords: mitochondria; brain; cognition; aging
MeSH Terms: conditions — Cognitive Dysfunction; Mental Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Novel nutritional product (containing Mitopure Urolithin A) targeting improvements in cognitive health
  Interventions: Dietary Supplement: Active Product
- Placebo (Placebo Comparator): Identical Placebo product
  Interventions: Dietary Supplement: Placebo Product

INTERVENTIONS:
Dietary Supplement: Active Product — Novel Nutritional Product targeting Cognition
  Arms: Active
Dietary Supplement: Placebo Product — Identical placebo product
  Arms: Placebo

SUMMARY:
This is a parallel group, randomized, double-blind, placebo-controlled clinical study assessing the safety and effects of a novel nutritional product on self-reported cognitive function and health in adults that reside in the USA. Participants will take their assigned study product (active or placebo) for 8 weeks and answer validated electronic surveys assessing cognitive function delivered to them through a text message (SMS) link or through email.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the following criteria:

* Adults, at least 40 years of age at the time of electronic consent, inclusive of all ethnicities, races, and gender identities

  o Assigned sex at birth will determine sex-specific recruitment and surveys (male vs female) employed, when needed
* Resides in the United States
* Has the opportunity for at least 30% improvement in their primary health outcome
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study

Exclusion Criteria:

Individuals who report any of the following during screening will be excluded from participation:

* Report being pregnant, trying to become pregnant, or breastfeeding
* Unable to provide a valid US shipping address and mobile phone number
* Reports current enrollment in another clinical trial
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English
* Reports a current and/or recent (up to 3 months ago) major illness and/or surgery that poses a known, significant safety risk.
* Reports a diagnosis of cardiac dysfunction, liver or kidney disease that presents a known contraindication and/or a significant safety risk with any of the study product ingredients.

  o NYHA Class III or IV congestive heart failure, atrial fibrillation, uncontrolled arrhythmias, cirrhosis, end-stage liver disease, stage 3b or 4 chronic kidney disease, or kidney failure
* Reports taking medications that have a well-established moderate or severe interaction, posing a substantial safety risk with any of the study product ingredients.

  o Anticoagulants, antihypertensives, anxiolytics, antidepressants, chemotherapy, immunotherapy, sedative hypnotics, seizure medications, medications that warn against grapefruit consumption, corticosteroids at doses greater than 5 mg per day, diabetic medications, oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection, antipsychotics, MAOIs, or thyroid products
* Reports current use of the primary ingredient(s) and/or similar product(s) to the active study product(s) that may limit the effects of the study products
* Lack of reliable daily access to the internet

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2025-07-29 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Cognitive function | 8 weeks
  Change in cognitive function score as assessed by PROMIS Cognitive Function 8A (scale 8-40; where higher scores correspond to better cognitive function)

SECONDARY OUTCOMES:
Fatigue | 8 weeks
  Change in fatigue score as assessed by Patient Reported Outcome Measurement System (PROMIS) Fatigue 4A (scale 4-20; where higher scores correspond to worse fatigue)
Sleep-related impairment | 8 weeks
  Change in sleep score as assessed by PROMIS Sleep-Related Impairment 4a (scale 4-20; where the higher scores correspond to worse sleep)
Cognitive abilities | 8 weeks
  Change in Cognitive Abilities score as assessed by PROMIS Cognitive Function - Abilities 8a (scale 8-40; where the higher scores correspond to better cognitive abilities)
Cognitive function (brain health) via smartphone application assessments | 8 weeks
  Change in cognitive function evaluated with DANA Brain Vital app
Minimal clinically important difference (MCID) in cognitive function | 8 weeks
  Likelihood of achieving minimal clinically important difference in cognitive function score as assessed by PROMIS Cognitive Function 8A (scale 8-40; where higher scores correspond to better cognitive function)
Minimal clinically important difference (MCID) in fatigue | 8 weeks
  Likelihood of achieving minimal clinically important difference in fatigue score as assessed by PROMIS Fatigue 4A (scale 4-20; where higher scores correspond to worse fatigue)
Minimal clinically important difference (MCID) in sleep | 8 weeks
  Likelihood of achieving minimal clinically important difference in sleep score, as measured by PROMIS Sleep-Related Impairment 4a (scale 4-20; where the higher scores correspond to worse sleep)
Minimal clinically important difference (MCID) in cognitive abilities | 8 weeks
  Likelihood of achieving minimal clinically important difference in cognitive abilities score as assessed by PROMIS Cognitive Function - Abilities 8a (scale 8-40; where the higher scores correspond to better cognitive abilities)
Adverse Events | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hewlings, PhD, Principal Investigator — Radicle Science Inc.
Locations (1):
- Radicle Science, Inc Office, Encinitas, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Radicle Science, Inc — https://radiclescience.com/